CLINICAL TRIAL: NCT06467890
Title: Knowledge of Vital Pulp Therapy in Permanent Teeth Among a Group of Dental Interns After Educational Programme: A Before and After Study
Brief Title: Knowledge of Vital Pulp Therapy in Permanent Teeth After Educational Programme: A Before and After Study
Status: Not yet recruiting | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mariam Maher Gindy, Teaching assistant in pediatric dentistry department, Cairo University
Other Study IDs: 69911
Record Dates: First submitted 2024-06-05; First posted 2024-06-21 (Actual); Last update posted 2024-06-21 (Actual); Status verified 2024-06

CONDITIONS: Pulp Disease, Dental; Knowledge
MeSH Terms: conditions — Dental Pulp Diseases

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Educational programme on vital pulp therapy: An educationnal programme based on the latest AAPD and AAE guidelines will be given to the participants after responding to the questionnaire for the first time.
  Interventions: Behavioral: Educational programme about vital pulp therapy

INTERVENTIONS:
Behavioral: Educational programme about vital pulp therapy — An awareness educational material based on the recent AAPD and AAE guidelines on vital pulp therapy will be sent to the participants right after they answer the questionnaire for the first time

SUMMARY:
evaluating the extent of knowledge of vital pulp therapy in permanent dentition among a group of dental interns in Egypt after educational programme.

DETAILED DESCRIPTION:
evaluating the extent of knowledge of vital pulp therapy in permanent dentition using a survey among a group of dental interns in Egypt after educational programme.

ELIGIBILITY:
Inclusion Criteria:

* Dental interns enrolled in the Pediatric Dentistry Department, Cairo University .
* Candidates who are willing to participate

Exclusion Criteria:

* Responses with incomplete information

Ages: 20 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Dental interns enrolled in the pediatric round in Cairo University
Sampling Method: Probability Sample
Enrollment: 550 (Estimated)
Dates: Start 2024-09-01 (Estimated); Primary Completion 2025-03-01 (Estimated); Study Completion 2025-05-30 (Estimated)

PRIMARY OUTCOMES:
Knowledge of vital pulp therapy | 6 months
  Online Questionnaire, percentage will be the measuring unit

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] AAE Position Statement on Vital Pulp Therapy. J Endod. 2021 Sep;47(9):1340-1344. doi: 10.1016/j.joen.2021.07.015. Epub 2021 Aug 3. No abstract available. PMID 34352305
- [Background] American Academy of Pediatric Dentistry. Pulp therapy for primary and immature permanent teeth. The Reference Manual of Pediatric Dentistry. Chicago, Ill.: American Academy of Pediatric Dentistry; 2022:415-23
- [Background] Bogen G, Dammaschke T, Chandler N. Vital pulp therapy. In: Berman L, Hargreaves KM, editors. Pathways of the Pulp. 12th ed. St. Louis, MO: Elsevier; 2021.
- [Background] Guan X, Zhou Y, Yang Q, Zhu T, Chen X, Deng S, Zhang D. Vital Pulp Therapy in Permanent Teeth with Irreversible Pulpitis Caused by Caries: A Prospective Cohort Study. J Pers Med. 2021 Nov 1;11(11):1125. doi: 10.3390/jpm11111125. PMID 34834477
- [Background] Parmar G, Singh S, Hegde JA, Kumar M, Kalyan S. Launching a new fellowship in microrestorative and endodontics for postgraduates in conservative dentistry and endodontics. J Conserv Dent. 2020 Jul-Aug;23(4):370-373. doi: 10.4103/JCD.JCD_328_20. Epub 2021 Jan 16. PMID 33623238
- [Background] Wisniewski JF, Norooz S, Callahan D, Mohajeri A. Survey of Vital Pulp Therapy Treatment in Permanent Dentition Being Taught at U.S. Dental Schools. J Endod. 2022 Sep;48(9):1107-1112. doi: 10.1016/j.joen.2022.06.009. Epub 2022 Jul 5. PMID 35798124
- [Background] Kakudate N, Yokoyama Y, Sumida F, Matsumoto Y, Gordan VV, Gilbert GH. Dentists' practice patterns of treatment for deep occlusal caries: Findings from a dental practice-based research network. J Dent. 2019 May;84:76-80. doi: 10.1016/j.jdent.2019.03.009. Epub 2019 Mar 29. PMID 30935965
- [Background] Doumani MD, Arnous WA, Alsafadi MF, Alnazer HA, Alanazi SM, Alotaibi KS, Al-Ammari AI. The Vital Pulp Therapy of Permanent Teeth: A Dental Practitioner's Perspective from Saudi Arabia. J Int Soc Prev Community Dent. 2020 Jun 15;10(3):300-308. doi: 10.4103/jispcd.JISPCD_69_19. eCollection 2020 May-Jun. PMID 32802776